CLINICAL TRIAL: NCT06981598
Title: Optimizing Psychological Health and Preventing Clinical Problems: Testing the Effectiveness of an Evidence-Based Toolkit for Integrated Operational Support
Brief Title: Prevention of Psychological Health Problems Via Integrated Operational Support
Acronym: IOS Toolkit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-FY2023-7921
Record Dates: First submitted 2025-03-17; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Depression, Anxiety; Grief; Leadership; Dissatisfaction
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Modified stepped wedge design training behavioral health technicians
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BH Technician Training (Experimental): BH Technician Training; active deliberate practice training
  Interventions: Behavioral: Cognitive Behavioral Coaching Training

INTERVENTIONS:
Behavioral: Cognitive Behavioral Coaching Training — Behavioral technicians will engage in a structured, deliberate-practice-based training program designed to enhance competence in evidence-based interventions (EBIs) over a 10-week period. The program begins with an initial seminar that provides an overview of the training framework, key research supporting deliberate practice, and specific intervention techniques. Each participant is assigned a coach-either a clinical psychologist or a licensed MSW with expertise in the EBI Toolkit-who will provide individualized guidance throughout the training. During the weekly coaching sessions, participants will review session notes, engage in structured practice exercises, and work toward mastering the skills and competencies necessary for effective intervention delivery. Weekly homework assignments will allow participants to practice each tool as though they were working with an SM client, followed by self-reflections that will be discussed in coaching sessions.

SUMMARY:
Sub-clinical behavioral health services in the military are performed by BH technicians, who receive minimal training. Due to this, embedding more technicians in military units is unlikely to benefit service members. Giving technicians training in, and access to, evidence-based interventions (EBI) could make their work more effective. The proposed study is a training trial examining the efficacy of the full integrated operational support (IOS) toolkit (evidence-based interventions for behavioral health), relative to routine care using standard resources, as a prevention resource for active-duty airmen.

DETAILED DESCRIPTION:
This study is conducted in collaboration with the Department of the Air Force (DAF) Medical Service to enhance the effectiveness of embedded behavioral health (BH) technicians in operational units. The initiative aligns with military health goals by embedding paraprofessional BH technicians within line units to improve service member (SM) access to mental health care, reduce stigma, and address risk factors such as sleep disorders, stress, trauma, and suicide prevention. However, variability in training and intervention delivery has limited their effectiveness. This research aims to test evidence-based training (EBT) approaches for BH technicians, equipping them with validated intervention tools and engagement techniques to improve SM psychological well-being, stress management, and service satisfaction.

The research builds on previous findings showing that embedded BH technicians increase accessibility and reduce stigma but often lack standardized training and structured intervention tools. The study will use a randomized controlled trial (RCT) design to compare trained vs. untrained BH technicians, assessing their adoption of evidence-based interventions (EBIs) and the resulting impact on SM well-being. The CBPR advisory board, which has guided the development of the IOS EBI Toolkit, will continue its role in refining training methods and implementation. Additionally, a patient advocate consultant, who has experienced suicidality, PTSD, and sleep disorders, will contribute to recruitment strategies and intervention refinement. This approach ensures that training is optimized for real-world military settings, increasing adoption and effectiveness.

The study's objectives are to evaluate whether EBI training improves BH technicians' adoption of intervention tools and SM outcomes, test whether BH technician competency mediates SM improvement, and deliver empirically supported training protocols to the DAF. The research aims to enhance the quality and impact of BH services in operational units, ultimately improving SM resilience, recovery, and mission readiness. By formalizing structured training programs and evidence-based engagement strategies, this initiative seeks to standardize and optimize the role of embedded BH technicians, ensuring they effectively support service members' mental health needs. If successful, these training protocols will be scaled for military-wide implementation, contributing to long-term mental health improvements across the DAF and broader military community.

ELIGIBILITY:
Inclusion Criteria:

* Service members seeing a behavioral health (BH) technician.
* Currently embedded BH technicians.

Exclusion Criteria:

* Service members who are not currently seeing a BH technician.
* BH technicians who are not embedded or have taken a clinic role.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5586 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Average Satisfaction of Service Members (SM) with Embedded Behavioral Health Technician (BHT) Services | From the SM's first session with their embedded BHT to their last session (up to 10 weeks)
  We will ask participating SMs questions about their session with their embedded BHT to gauge their satisfaction with the experience. The questions are prompts such as "How much do you think your meeting today will help you deal with your current difficulties?" and How much do you think working with a MHT/BHT/psych/4C will help you improve the things you would like to change?"
Change in Service Member PHQ-9 (Patient Health Questionnaire-9) Score | From the SM's first session with their embedded BHT to one month after their last session with their embedded BHT (up to 14 months after the completion of the baseline survey after the first appointment with their embedded BHT)
  The PHQ-9 (Patient Health Questionnaire-9) measures physical, emotional, and cognitive symptoms of Major Depression such as "feeling down, depressed, or hopeless," "trouble falling or staying asleep, or sleeping too much," or "trouble concentrating on things, such as reading the newspaper or watching television." Service members (SM) will fill out this measure.
Change in Service Member WHO-5 Well-being Index Score | From the SM's first session with their embedded BHT to one month after their last session with their embedded BHT (up to 14 months after the completion of the baseline survey after the first appointment with their embedded BHT)
  The WHO-5 Well-being Index measures general well-being with prompts such as "I have felt cheerful and in good spirits" and "I woke up feeling fresh and rested." Service members (SM) will fill out this measure.
Change in Service Member PSS-10 (Perceived Stress Scale - 10 item version) Score | From the SM's first session with their embedded BHT to one month after their last session with their embedded BHT (up to 14 months after the completion of the baseline survey after the first appointment with their embedded BHT)
  The PSS-10 (Perceived Stress Scale - 10 item version) measures the SM's stress with prompts such as: "In the last month, how often have you felt that you were unable to control the important things in your life?" and "In the last month, how often have you felt that you were on top of things?" Service members (SM) will fill out this measure.
Change in Service Member STAI (State-Trait Anxiety Inventory) Score | From the SM's first session with their embedded BHT to one month after their last session with their embedded BHT (up to 14 months after the completion of the baseline survey after the first appointment with their embedded BHT)
  The STAI (State-Trait Anxiety Inventory) measures anxiety by asking participants about their current emotions with prompts such as "I feel calm," "I feel frightened," and "I feel nervous." Service members (SM) will fill out this measure.

SECONDARY OUTCOMES:
Frequency of evidence based intervention (EBI) use among behavioral health technicians (BHT) following IOS Toolkit Cognitive Behavioral Coaching training | Pre-training (10-week period) to post-training (10-week period)
  The percentage of all interventions offered by BHTs while treating service members that are evidence based will be compared to the percentage that are not evidence based from pre-training (10-week period) to post-training (10-week period).

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Slep, PhD, Principal Investigator — NYU
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No